CLINICAL TRIAL: NCT02547311
Title: Shared Medical Appointments to Improve Outcomes in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-1281; #2015PG-T1D080 (Other: UCDenver)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Team Clinic Intervention (Experimental): Middle School and High School Team Clinic Intervention
  Interventions: Behavioral: Team Clinic
- Standard Clinical Care - Control (No Intervention): Standard Clinical Care - Control

INTERVENTIONS:
Behavioral: Team Clinic
  Arms: Team Clinic Intervention

SUMMARY:
Adolescents and emerging adults with type 1 diabetes (T1D) experience significant struggles with their diabetes management resulting in worsening diabetes health and increased complications. This population's declining well-being occurs during a time when they should be at their healthiest and enjoying multiple exciting life transitions. Their worsening diabetes management is complicated by the fact they are also learning how to become more independent from their family in preparation for eventually leaving home. Furthermore, the number of people under 20 years of age diagnosed with T1D has increased dramatically over the past 10 years giving rise to increased concern about providing care to this population.

The Team Clinic Intervention is an innovative clinical care approach to address the medical and developmental needs of adolescents with T1D and their families. A group medical appointment format will be used for routine diabetes clinic visits in middle school and high school adolescents with T1D. Parents of these patients will be participating in their own group during these clinic visits. The Team Clinic model incorporates developmentally tailored peer support and novel learning tools, (e.g. games, physical activity, and/or interaction through Internet resources, e.g. blogs, forums) into the shared medical appointment design.

The goal of Team Clinic Intervention is to improve medical and psychological outcomes in adolescents with T1D and their parents. The study will investigate, in a randomized controlled trial, the efficacy of a novel clinical care model that addresses the unique developmental strengths and weaknesses of the T1D adolescent population. The Team Clinic format streamlines clinical care delivery to this often-challenging patient population without placing additional burden on youth, families, or clinics because the intervention will be completed during routine diabetes care visits. Moreover, the Team Clinic approach maximizes the benefits of peer support by delivering care in a group format to address the sense of isolation that teens and families coping with chronic illness often feel.

If successful, the Team Clinic Intervention will not only positively impact adolescents with T1D and their families, but it could be used as a model of care for other adolescents with chronic medical conditions struggling to remain involved and invested in their medical care. Team Clinics may be one approach to successfully engaging adolescents in their diabetes care prior to their transition away from home, which will help them remain invested and active in their medical care through adolescence and young adulthood.

ELIGIBILITY:
Inclusion Criteria:

* T1D >1 year duration, 6th-10th grade

Exclusion Criteria:

* non-English speaking
* severe behavioral, developmental, or psychological diagnosis making group participation difficult

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 30 months
  Hemoglobin A1c
Satisfaction Questionnaire | 30 months
  Clinic satisfaction (patient and parent)
Diabetes distress Questionnaire | 30 months
  Diabetes distress (patient and parent)
Cost effectiveness | 30 months
  Clinical cost effectiveness of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Raymond, MD, MCR, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver School of Medicine Barbara Davis Center, Aurora, Colorado, United States